CLINICAL TRIAL: NCT02568449
Title: A Phase II Trial of BIBF 1120 (Nintedanib) in Recurrent Malignant Pleural Mesothelioma
Brief Title: Nintedanib in Treating Patients With Malignant Pleural Mesothelioma That Is Recurrent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dipesh Uprety, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-010; NCI-2015-01412 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1506014121; 2015-010 (Other: Wayne State University/Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Recurrent Pleural Malignant Mesothelioma; Stage IV Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nintedanib) (Experimental): Patients receive nintedanib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Given PO
  Other Names: BIBF 1120; BIBF-1120; Intedanib; Multitargeted Tyrosine Kinase Inhibitor BIBF 1120; tyrosine kinase inhibitor BIBF 1120; Vargatef

SUMMARY:
This phase II trial studies how well nintedanib works in treating patients with malignant pleural mesothelioma that has come back. Nintedanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the 4-month progression-free survival (PFS) in patients with recurrent, unresectable malignant pleural mesothelioma (MAM) treated with nintedanib.

SECONDARY OBJECTIVES:

I. To assess response rate (confirmed and unconfirmed, complete and partial responses) and disease control rate (response or stable disease) in the subset of patients with measurable disease by both RECIST (Response Evaluation Criteria in Solid Tumors) 1.1 criteria and Modified RECIST criteria for pleural tumors.

II. To assess overall survival.

III. To evaluate the frequency and severity of toxicities associated with this treatment regimen.

IV. To collect tissue samples for future correlative studies related to overall study objectives.

OUTLINE:

Patients receive nintedanib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of unresectable malignant pleural mesothelioma
* Patients must have measurable or non-measurable disease documented by computed tomography (CT) scan; measurable disease must be assessed within 28 days prior to registration; non-measurable disease must be assessed within 42 days prior to registration; the CT from a combined positron emission tomography (PET)/CT must not be used to document measurable disease unless it is of diagnostic quality; all disease must be assessed by RECIST and modified RECIST criteria
* Patients must have had prior systemically administered platinum-based chemotherapy; pleural space washing with cisplatin does not constitute systemic administration; no more than two prior systemic therapeutic regimens are allowed (including biologics, targeted and immunotherapies), and at least one regimen must have been platinum-based; neoadjuvant and/or adjuvant systemic therapy will not be counted as a prior regimen, assuming at least 12 weeks have elapsed between the end of neoadjuvant/adjuvant therapy and development of progressive disease; patients must have completed systemic therapy (including any chemotherapy, biologics, targeted and immunotherapies) >= 28 days (42 days for nitrosoureas or mitomycin C) prior to registration and have recovered from adverse events due to agents administered
* No prior treatment with BIBF 1120 or any other vascular endothelial growth factor receptor (VEGFR) inhibitor
* No known hypersensitivity to BIBF 1120, to its excipients or to contrast media
* Patients may have received prior surgery (e.g., pleurectomy) provided that at least 28 days have elapsed since surgery (thoracic or other major surgeries) and patients have recovered from all associated toxicities at the time of registration; there must be no anticipated need for major surgical procedures during protocol treatment
* No active brain metastases (e.g. stable for < 4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anti-convulsants; dexamethasone therapy will be allowed if administered as stable dose for at least one month before randomization); no leptomeningeal disease
* No radiographic evidence of cavitary or necrotic tumors
* No centrally located tumors with radiographic evidence (CT or magnetic resonance imaging [MRI]) of local invasion of major blood vessels
* Institutions must offer patients the opportunity to submit tissue for future correlative studies
* Patients may have received prior radiation therapy provided that at least 14 days have elapsed since the last treatment and patients have recovered from all associated toxicities at the time of registration
* Patients must have a Zubrod performance status of 0-1
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Platelet count >= 100,000/mcl
* Serum bilirubin =< institutional upper limit of normal (IULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) must be =< 1.5 x IULN; for patients with liver metastasis, NO total bilirubin outside of normal limits, and NO ALT or AST > 2.5 ULN
* Serum creatinine =< 1.5 x IULN or a calculated or measured creatinine clearance >= 50 mL/min using the following formula: calculated creatinine clearance = (140-age) x wt (weight) (kg) x 0.85 (if female)/72 x creatinine (mg/dl); these tests (including creatinine [mg/dl] if using calculated creatinine clearance) must be obtained within 14 days prior to registration
* No proteinuria Common Terminology Criteria For Adverse Events (CTCAE) grade 2 or greater
* No therapeutic anticoagulation (except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous device) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid < 325mg per day); no history of clinically significant haemorrhagic or thromboembolic event in the past 6 months
* Patients must have no evidence of bleeding diathesis or coagulopathy; patients must have no pathologic condition other than mesothelioma that carries a high risk of bleeding
* No major injuries within the past 10 days prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period
* Patients must not have gastrointestinal tract disease resulting in an inability to take oral or enteral medication via a feeding tube or a requirement for intravenously (IV) alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease
* No significant cardiovascular diseases ( i.e. uncontrolled hypertension, unstable angina, history of infarction within the past 12 months prior to start of study treatment, congestive heart failure > NYHA [New York Heart Association Class] II, serious cardiac arrhythmia, pericardial effusion)
* No active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy
* No active or chronic hepatitis C and/or B infection
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* No psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule
* No active alcohol or drug abuse
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dipesh Uprety, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (3):
- United States (3):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nintedanib)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 16
Age, Continuous [Median (Full Range); unit: years] | 70 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS will be estimated using standard Kaplan-Meier methods for censored data, from which the median and other statistics of interest will be calculated (e.g., rates at 3 months, 6 months, 12 months).
Time Frame: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause; assessed up to 4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 20
months | 1.8 [1.5 to 3.5]

2. Secondary Outcome: Incidence of Grade 3-4 Toxicity
Description: Number of participants with grade 3 or grade 4 for each type of toxicity encountered, using all toxicity evaluable patients.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 20
Participants
  Dyspnea (shortness of breath) | 5
  Lymphopenia | 4
  Hypoxia | 2
  Syncope (fainting) | 1
  pulmonary/upper respiratory- other, acute respiratory event | 1
  Thrombosis/thrombus/embolism | 1
  Encephalopathy | 1
  Pericardial effusion | 1
  Pain - Chest wall | 1
  Ascites (non-malignant) | 1
  Edema: trunk/genital | 1
  Supraventricular and nodal arrhythmia - Atrial fibrillation | 1

3. Secondary Outcome: Overall Survival
Description: Overall survival will be estimated using standard Kaplan-Meier methods for censored data, from which the median and other statistics of interest will be calculated (e.g., rates at 3 months, 6 months, 12 months).
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 20
months | 4.1 [2.5 to 8.7]

4. Secondary Outcome: Number of Participants Responded (Complete Response, Partial Response, Stable Disease, Progressive Disease, Not Evaluable)
Description: number of participants responded (complete response, partial response, stable disease, progressive disease, not evaluable) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0)
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 20
Participants
  complete response | 0
  partial response | 0
  stable disease | 0
  progressive disease | 18
  not evaluable | 2

ADVERSE EVENTS:
Time Frame: Up to one year.
Arm/Group | Treatment (Nintedanib)
All-Cause Mortality (participants affected / at risk) | 15/20
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nintedanib) (N=20)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4)
Syncope (fainting) (Nervous system disorders) | 1 (1)
pulmonary/upper respiratory- other, acute respiratory event (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Edema: trunk/genital (Blood and lymphatic system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nintedanib) (N=20)
ALT, SGPT (Blood and lymphatic system disorders) | 3 (3)
AST, SGOT (Blood and lymphatic system disorders) | 6 (6)
Albumin, serum-low (hypoalbuminemia) (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Ascites (non-malignant) (Gastrointestinal disorders) | 2 (2)
Calcium, serum-low (hypocalcemia) (Blood and lymphatic system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Creatinine (Blood and lymphatic system disorders) | 7 (7)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 17 (17)
Distension/bloating, abdominal (Gastrointestinal disorders) | 3 (3)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Edema: limb (Blood and lymphatic system disorders) | 7 (7)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 13 (13)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 2 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 11 (11)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5)
Hypertension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4)
Magnesium, serum-low (hypomagnesemia) (Blood and lymphatic system disorders) | 3 (3)
Mood alteration - Anxiety (Nervous system disorders) | 2 (2)
Nausea (General disorders) | 4 (4)
Pain - Abdomen NOS (General disorders) | 7 (7)
Pain - Chest wall (General disorders) | 6 (6)
Pain - Chest/thorax NOS (General disorders) | 2 (2)
Pain - Head/headache (General disorders) | 2 (2)
Pain - Other (Specify, __) (General disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 3 (3)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Potassium, serum-high (hyperkalemia) (Blood and lymphatic system disorders) | 6 (6)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No